CLINICAL TRIAL: NCT00983476
Title: Web-Based Delivery of MOVE! to Veterans With Serious Mental Illness
Brief Title: Web-Based Delivery of MOVE! to Veterans With Serious Mental Illness (SMI)
Acronym: Web-MOVE!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 09-083
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Psychotic Disorders; Obesity; Health Behaviors
Keywords: Randomized controlled trial; Obesity; Comparative Effectiveness; Clinical practice guidelines; Medical Informatics Computing; Services, Mental Health; Self-care; Psychotic disorders; Mental Health Care; Veterans
MeSH Terms: conditions — Psychotic Disorders; Obesity; Health Behavior; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): in-person MOVE! SMI
  Interventions: Behavioral: in-person MOVE! SMI
- Arm 2 (Experimental): web-based MOVE! SMI
  Interventions: Behavioral: web-based MOVE! SMI
- Arm 3 (No Intervention): usual care + educational handouts regarding weight loss

INTERVENTIONS:
Behavioral: in-person MOVE! SMI — Individual and group in-person sessions that deliver manualized MOVE! curriculum adapted for use with individuals with cognitive deficits (often found in individuals with severe mental illness (SMI))
  Arms: Arm 1
Behavioral: web-based MOVE! SMI — online sessions that deliver manualized MOVE! curriculum adapted for use with individuals with cognitive deficits (often found in individuals with severe mental illness (SMI))
  Arms: Arm 2

SUMMARY:
Obesity and physical inactivity have reached epidemic proportions, resulting in increased rates of a variety of chronic diseases, increased risk of death, and substantial health care costs. Individuals with serious mental illness are even more likely to be overweight or obese, which contributes to the high rate of co-morbid medical disease and early mortality found among this population. Specific individual and group-based psychoeducational interventions have repeatedly and consistently been shown to help adults with serious mental illness improve their weight. However, these require substantial time from mental health clinicians, and frequent visits by patients to mental health clinics. This creates challenges for patients who may need to travel to a medical center that provides these services, and who often have limited transportation options. It is likely that these barriers can be addressed with a computerized, web-based intervention focused on diet and exercise education, and tailored for veterans with serious mental illness. Web-based systems can deliver content that is intensive, engaging, and tailored to the needs and preferences of specific patients. Web-based systems can be delivered using computers at community-based outpatient Clinics or other settings in the community. The objective of this project is to develop and evaluate the effectiveness of a web-based intervention to help patients with serious mental illness lose weight.

DETAILED DESCRIPTION:
Background: Obesity has reached epidemic proportions, and often has serious adverse health consequences. The VA has deployed a "MOVE! Weight Management Program" nationally in the general patient population. Since individuals with serious mental illness (SMI) often have cognitive deficits, specialized psychoeducational interventions are needed in this population. Specialized psychoeducational interventions for weight have been developed and studied in populations with SMI. This evidence-based practice has been adapted for use in VA, resulting in a "MOVE! SMI" intervention. However, it has proven to be quite difficult to disseminate this intervention. Patients with SMI often have limited transportation options, and may not want to participate in groups. Also, in-person MOVE! SMI requires substantial time from mental health clinicians. This clinician time has been difficult to deploy or is not available at many clinic locations. It is likely that these barriers can be addressed with a computerized, web-based version of MOVE! . Specialized web-based approaches have been studied and found to be successful in people with SMI, and can deliver content that is intensive and engaging with minimal requirements for staff time.

Objectives: The VA Network 5 and 22 Mental Illness Research, Education, and Clinical Centers (MIRECCs) developed a web-based system that provides computerized counseling regarding diet to individuals with SMI. The proposed project expanded this system. This project's objectives are to: 1) develop a comprehensive web-based system that delivers MOVE! using design features that meet the needs of individuals with mental illness; 2) evaluate the effectiveness, in patients with serious mental illness, of web-based MOVE! compared with in-person MOVE! and a control group; and, 3) characterize, from the patient's perspective, the strengths, weaknesses, and barriers to the use of in-person and web-based MOVE!.

Methods: This is a prospective, randomized, controlled trial in patients with SMI who are obese and receiving treatment with medications that often have weight gain as a major side-effect. Participants are assigned to in-person MOVE! SMI, web-based MOVE! SMI with support from peer coaches, or a comparison group. Research assessments occur at 0, 3, 6, 9 and 12 months. Changes in outcomes are compared over time between the three groups. Comparative effectiveness is evaluated at 6 months. A secondary objective is to evaluate the extent to which gains are maintained at 9 and 12 months.

Status: The project team developed the needed materials, methods, and informatics systems. Patients were enrolled, and study enrollment and interventions are complete. Follow up interviews are complete and the interventions have been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual (DSM-IV) diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, recurrent major depressive disorder with psychosis, or PTSD;
* age 18 and over;
* no psychiatric hospitalization during the month prior to enrollment;
* receipt of an antipsychotic medication for at least 3 months prior to enrollment;
* BMI of 30 or higher, or BMI of 28 or higher if 10 pounds of recent weight gain;
* medical clearance to participate from a VA physician;
* control over diet.

Exclusion Criteria:

* any medical condition for which a weight program is contraindicated;
* history of bariatric surgery;
* pregnant and nursing mothers;
* a diagnosis of dementia;
* not able to provide informed consent by self or legally appointed representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2012-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander S Young, MD MSHS, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cohen AN, Golden JF, Young AS. Peer wellness coaches for adults with mental illness. Psychiatr Serv. 2014 Jan 1;65(1):129-30. doi: 10.1176/appi.ps.650101. No abstract available. PMID 24382767
- [Derived] Muralidharan A, Brown CH, Zhang Y, Niv N, Cohen AN, Kreyenbuhl J, Oberman RS, Goldberg RW, Young AS. Quality of life outcomes of web-based and in-person weight management for adults with serious mental illness. J Behav Med. 2020 Oct;43(5):865-872. doi: 10.1007/s10865-019-00117-1. Epub 2019 Nov 18. PMID 31741204
- See also: VA MOVE! Program — http://www.move.va.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2012 and April 2014, we obtained a list of individuals at the study site who met inclusion criteria for psychiatric diagnosis, age, and psychotropic medication. Study flyers were also posted in mental health clinics. 1429 individuals were screened for eligibility, and 19% were eligible, interested, enrolled, and randomized.
Pre-assignment Details: 7 patients were withdrawn by the PI when they were determined to be ineligible, after signing a consent. Ineligibility reasons included: not being prescribed inclusion criteria medication, not receiving approval from primary care physician, non-veteran status, and unable to consent to participation. 2 patients disenrolled prior to group assignment.
Groups:
- Arm 1: In-person MOVE! SMI: In-person MOVE! SMI: Individual and group in-person sessions that deliver manualized MOVE! diet and activity curriculum adapted for use with individuals with severe mental illness (SMI), who often have cognitive deficits
- Arm 2: Web-based MOVE! SMI: Web-based MOVE! SMI: online sessions that deliver manualized MOVE! diet and activity curriculum adapted for use with individuals with severe mental illness (SMI), who often have cognitive deficits; plus peer coaching
- Arm 3: Usual Care + Handouts: usual care + educational handouts regarding weight loss
Period: Overall Study
Arm/Group | Arm 1: In-person MOVE! SMI | Arm 2: Web-based MOVE! SMI | Arm 3: Usual Care + Handouts
Started | 95 | 93 | 88
6 Month Follow up Assessment | 71 | 62 | 74
Completed | 78 | 71 | 88
Not Completed | 17 | 22 | 0
Not completed — Did not receive intervention | 17 | 22 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: In-person MOVE! SMI: in-person MOVE! SMI
  in-person MOVE! SMI: Individual and group in-person sessions the deliver manualized MOVE! curriculum adapted for use with individuals with cognitive deficits (often found in individuals with severe mental illness (SMI))
- Arm 2: Web-based MOVE! SMI: web-based MOVE! SMI
  web-based MOVE! SMI: online sessions the deliver manualized MOVE! curriculum adapted for use with individuals with cognitive deficits (often found in individuals with severe mental illness (SMI))
- Total: Total of all reporting groups
Arm/Group | Arm 1: In-person MOVE! SMI | Arm 2: Web-based MOVE! SMI | Arm 3: Usual Care + Handouts | Total
Number analyzed (Participants) | 95 | 93 | 88 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (9.6) | 54.7 (8.9) | 54.2 (9.9) | 54.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Observation of gender as male or female
  Participants
    Female | 7 | 8 | 2 | 17
    Male | 88 | 85 | 86 | 259
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 5 | 1 | 7
  Asian | 3 | 0 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
  Black or African American | 43 | 43 | 45 | 131
  White | 36 | 35 | 32 | 103
  More than one race | 5 | 3 | 3 | 11
  Unknown or Not Reported | 7 | 7 | 3 | 17
Education [Number; unit: participants] — Patient reported educational level
  participants
    High School, no diploma | 5 | 2 | 6 | 13
    High School diploma or some college | 60 | 64 | 56 | 180
    Degree (2 or 4 year) | 27 | 24 | 22 | 73
    Graduate School (Degree or no degree) | 3 | 3 | 4 | 10
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/(meters squared)] — BMI = (weight in pounds * 703)/ height in inches²
  kg/(meters squared) | 34.9 (5.0) | 34.2 (5.3) | 34.4 (5.6) | 34.5 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index (BMI)
Description: BMI = (weight in pounds * 703)/ (height in inches²) at 6 month follow-up as predicted by the mixed model described in Statistical Analysis 1
Time Frame: 6 months
Population: All randomized participants who received any intervention as randomized were included in the primary analyses, regardless of the number of assessments completed. Receiving intervention as randomized was defined as participating in one or more modules/sessions (WebMOVE or MOVE SMI) or receipt of the educational handout (Usual Care).
Measure: Mean (Standard Error); unit: kg/(meters squared)
Groups:
- Arm 1: In-person MOVE! SMI: Individual and group in-person sessions that deliver manualized MOVE! curriculum adapted for use with individuals with cognitive deficits (often found in individuals with severe mental illness (SMI))
- Arm 2: Web-based MOVE! SMI: online sessions that deliver manualized MOVE! curriculum adapted for use with individuals with cognitive deficits (often found in individuals with severe mental illness (SMI))
Arm/Group | Arm 1: In-person MOVE! SMI | Arm 2: Web-based MOVE! SMI | Arm 3: Usual Care + Handouts
Number analyzed (Participants) | 78 | 71 | 88
kg/(meters squared) | 34.9 (0.4) | 33.4 (0.4) | 34.4 (0.4)
Statistical Analysis 1: Comparison: Arm 1: In-person MOVE! SMI vs Arm 2: Web-based MOVE! SMI vs Arm 3: Usual Care + Handouts; Difference in Body Mass Index (BMI) by study arm at 6 months after controlling for BMI 6 months prior to baseline using a repeated measures mixed model with arm, time, and the interaction of arm by time; Test type: Superiority or Other; p = 0.11, Mixed Models Analysis; Slope = 2.2 — Reference group is Web-based MOVE SMI: In-person MOVE SMI visit x group Beta estimate is .27 (p=.08); Reference group is Web-based MOVE SMI: Usual care plus handouts visit x group Beta estimate is .29 (p=.06)

2. Primary Outcome: Body Mass Index (BMI) Within Obese Sample
Description: BMI = (weight in pounds * 703)/ (height in inches²); obese defined as BMI > 30
Time Frame: 6 months
Population: Analyses excluded participants with BMI of 28-29.9 (overweight) at baseline, leaving only those with BMI >= 30 at baseline who received the intervention as randomized.
Measure: Mean (Standard Error); unit: kilogram/(meters squared)
Groups:
- Arm 1: In-person MOVE! SMI: Individual and group in-person sessions that deliver manualized MOVE! diet and activity curriculum adapted for use with individuals with severe mental illness (SMI), who often have cognitive deficits
- Arm 2: Web-based MOVE! SMI: online sessions that deliver manualized MOVE! diet and activity curriculum adapted for use with individuals with severe mental illness (SMI), who often have cognitive deficits; plus peer coaching
Arm/Group | Arm 1: In-person MOVE! SMI | Arm 2: Web-based MOVE! SMI | Arm 3: Usual Care + Handouts
Number analyzed (Participants) | 68 | 59 | 73
kilogram/(meters squared) | 35.9 (0.4) | 34.2 (0.4) | 35.6 (0.4)
Statistical Analysis 1: Comparison: Arm 1: In-person MOVE! SMI vs Arm 2: Web-based MOVE! SMI vs Arm 3: Usual Care + Handouts; In the obese sample, difference in Body Mass Index (BMI) by study arm at 6 months after controlling for BMI 6 months prior to baseline using a repeated measures mixed model with arm, time, and the interaction of arm by time; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Slope = 4.02 — Reference group is Web-based MOVE SMI: In-person MOVE SMI visit x group Beta estimate is .40 (p=.02); Reference group is Web-based MOVE SMI: Usual care plus handouts visit x group Beta estimate is .44 (p=.01)

3. Primary Outcome: Dietary Habits: Reducing Calories (Self-efficacy, Motivation, Readiness to Change)
Description: Self-Efficacy and Eating Habits Survey (Sallis et al., 1988): Reducing Calories Factor.
  The Reducing Calories factor includes survey items 6-10, which are each scored on a scale from 1-5. The factor score is an average of the scores on those items. Higher scores indicate more confidence in making the change in reducing calories. Range in the factor scores can be from 1 (min) to 5 (max).
Time Frame: 6 months
Population: All randomized participants who received the intervention as randomized and completed this measure at 6 months were included in the analysis. Receiving the intervention as randomized was minimally defined as participating in one or more modules/sessions (WebMOVE or MOVE SMI) or receipt of the educational handout (Usual Care).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1: In-person MOVE! SMI | Arm 2: Web-based MOVE! SMI | Arm 3: Usual Care + Handouts
Number analyzed (Participants) | 68 | 61 | 74
units on a scale | 4.1 (0.11) | 3.9 (0.11) | 4.0 (0.10)
Statistical Analysis 1: Comparison: Arm 1: In-person MOVE! SMI vs Arm 2: Web-based MOVE! SMI vs Arm 3: Usual Care + Handouts; Test type: Superiority or Other; p = 0.32, ANOVA; Mean Difference (Final Values) = 1.14 — No comparison between groups was conducted because overall model test was not statistically significant

4. Primary Outcome: Dietary Habits: Reducing Fat (Self-efficacy, Motivation, Readiness to Change)
Description: Self-Efficacy and Eating Habits Survey (Sallis et al., 1988): Reducing Fat Factor.
  The Reducing Fat factor includes survey items 16-20, which are each scored on a scale from 1-5. The factor score is an average of the scores on those items. Higher scores indicate more confidence in making the change in reducing fat in the diet. Range in the factor scores can be from 1 (min) to 5 (max).
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1: In-person MOVE! SMI | Arm 2: Web-based MOVE! SMI | Arm 3: Usual Care + Handouts
Number analyzed (Participants) | 68 | 61 | 74
units on a scale | 4.1 (0.11) | 3.9 (0.11) | 3.8 (0.11)
Statistical Analysis 1: Comparison: Arm 1: In-person MOVE! SMI vs Arm 2: Web-based MOVE! SMI vs Arm 3: Usual Care + Handouts; Test type: Superiority or Other; p = 0.11, ANOVA; Mean Difference (Final Values) = 2.23 — No comparison between groups was conducted because overall model test was NS

5. Secondary Outcome: Quality of Life: Physical Functioning
Description: Impact of Weight on Quality of Life (IWQOL; Kolotkin et al., 2008): Physical Functioning subscale.
  The Physical Functioning subscale includes survey items 1-11, which are each scored on a scale from 1-5. The subscale score is an average of the scores on those items. Lower scores indicate greater impairment. Range in the subscale scores can be from 1 (min) to 5 (max).
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Arm 1: In-person MOVE! SMI: Individual and group in-person sessions the deliver manualized MOVE! curriculum adapted for use with individuals with cognitive deficits (often found in individuals with severe mental illness (SMI))
- Arm 2: Web-based MOVE! SMI: online sessions the deliver manualized MOVE! curriculum adapted for use with individuals with cognitive deficits (often found in individuals with severe mental illness (SMI))
Arm/Group | Arm 1: In-person MOVE! SMI | Arm 2: Web-based MOVE! SMI | Arm 3: Usual Care + Handouts
Number analyzed (Participants) | 68 | 61 | 74
units on a scale | 2.4 (0.1) | 2.4 (0.1) | 2.6 (0.1)
Statistical Analysis 1: Comparison: Arm 1: In-person MOVE! SMI vs Arm 2: Web-based MOVE! SMI vs Arm 3: Usual Care + Handouts; Test type: Superiority or Other; p = 0.47, ANOVA; Mean Difference (Final Values) = 0.75 — No comparison between groups was conducted because overall model test was NS

6. Secondary Outcome: Quality of Life: Self-Esteem
Description: Impact of Weight on Quality of Life (IWQOL; Kolotkin et al. 2008): Self-Esteem subscale.
  The Self-Esteem subscale includes survey items 12-18, which are each scored on a scale from 1-5. The subscale score is an average of the scores on those items. Lower scores indicate greater impairment. Range in the subscale scores can be from 1 (min) to 5 (max).
Time Frame: 6 months
Population: All randomized participants who received the intervention as randomized and had data at 6 months were included in the analyses. Receiving the intervention as randomized was minimally defined as participating in one or more modules/sessions (WebMOVE or MOVE SMI) or receipt of the educational handout (Usual Care).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1: In-person MOVE! SMI | Arm 2: Web-based MOVE! SMI | Arm 3: Usual Care + Handouts
Number analyzed (Participants) | 68 | 61 | 74
units on a scale | 2.3 (0.13) | 2.3 (0.14) | 2.5 (0.13)
Statistical Analysis 1: Comparison: Arm 1: In-person MOVE! SMI vs Arm 2: Web-based MOVE! SMI vs Arm 3: Usual Care + Handouts; Test type: Superiority or Other; p = 0.51, ANOVA; Mean Difference (Final Values) = 0.67 — No comparison between groups was conducted because overall model test was NS

7. Secondary Outcome: Quality of Life: Sexual Life
Description: Impact of Weight on Quality of Life (IWQOL; Kolotkin et al 2008): Sexual Life subscale.
  The Sexual Life subscale includes survey items 19-22, which are each scored on a scale from 1-5. The subscale score is an average of the scores on those items. Lower scores indicate greater impairment. Range in the subscale scores can be from 1 (min) to 5 (max).
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1: In-person MOVE! SMI | Arm 2: Web-based MOVE! SMI | Arm 3: Usual Care + Handouts
Number analyzed (Participants) | 67 | 61 | 74
units on a scale | 1.7 (0.12) | 1.8 (0.13) | 1.7 (0.11)
Statistical Analysis 1: Comparison: Arm 1: In-person MOVE! SMI vs Arm 2: Web-based MOVE! SMI vs Arm 3: Usual Care + Handouts; Test type: Superiority or Other; p = 0.83, ANOVA; Mean Difference (Final Values) = 0.19 — No comparison between groups was conducted because overall model test was NS

8. Secondary Outcome: BMI
Description: BMI = (weight in pounds * 703)/ height in inches²
Time Frame: 9 months
Population: All randomized participants who received the intervention as randomized and who completed a 9 month follow-up weight were included in this summary. Receiving the intervention as randomized was minimally defined as participating in one or more modules/sessions (WebMOVE or MOVE SMI) or receipt of the educational handout (Usual Care).
Measure: Mean (Standard Deviation); unit: kg/meter squared
Groups:
- Arm 1: In-person MOVE! SMI: in-person MOVE! SMI
  in-person MOVE! SMI: Individual and group in-person sessions that deliver manualized MOVE! curriculum adapted for use with individuals with cognitive deficits (often found in individuals with severe mental illness (SMI))
- Arm 2: Web-based MOVE! SMI: web-based MOVE! SMI
  web-based MOVE! SMI: online sessions that deliver manualized MOVE! curriculum adapted for use with individuals with cognitive deficits (often found in individuals with severe mental illness (SMI))
Arm/Group | Arm 1: In-person MOVE! SMI | Arm 2: Web-based MOVE! SMI | Arm 3: Usual Care + Handouts
Number analyzed (Participants) | 60 | 55 | 69
kg/meter squared | 34.9 (6.0) | 33.0 (4.8) | 34.2 (6.1)

9. Secondary Outcome: BMI
Description: BMI = (weight in pounds * 703)/ height in inches²
Time Frame: 12 months
Population: All randomized participants who received the intervention as randomized and who completed a 12 month follow-up weight were included in this summary. Receiving the intervention as randomized was minimally defined as participating in one or more modules/sessions (WebMOVE or MOVE SMI) or receipt of the educational handout (Usual Care).
Measure: Mean (Standard Deviation); unit: kg/meter square
Arm/Group | Arm 1: In-person MOVE! SMI | Arm 2: Web-based MOVE! SMI | Arm 3: Usual Care + Handouts
Number analyzed (Participants) | 62 | 58 | 76
kg/meter square | 34.7 (6.6) | 32.4 (4.9) | 34.0 (6.2)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for a period of 3 years, from the start of recruitment in 2012 through the completion of all data collection in 2015.
Description: Adverse events were likely not related to the interventions or the study and therefore were not further categorized beyond the outcome of the event (i.e., hospitalization, death).
Arm/Group | Arm 1: In-person MOVE! SMI | Arm 2: Web-based MOVE! SMI | Arm 3: Usual Care + Handouts
Serious Adverse Events (participants affected / at risk) | 1/95 | 2/93 | 2/88
Other Adverse Events (participants affected / at risk) | 0/95 | 0/93 | 0/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: In-person MOVE! SMI (N=95) | Arm 2: Web-based MOVE! SMI (N=93) | Arm 3: Usual Care + Handouts (N=88)
Patient death (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — On 08/13/2012 while attempting to reach the patient for f/u interview, research staff was notified that the patient died on 7/25/12. This Event is anticipated in this population, and was unrelated to the study (heart failure).
Hospitalization (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Subject was meeting with study staff and mentioned that he had been experiencing chest pain since the previous night. Staff escorted subject to main hospital for assessment, where he was later admitted.
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Subject's psychiatrist informed research staff that subject was admitted for psychiatric stabilization, as he has been poorly adherent to his psychiatric medication regimen and demonstrating increasingly inappropriate behaviors.
Patient death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — On 1/14/14 while attempting to reach the patient for f/u interview, research staff was notified by the patient's sister that he died "around Christmas". This adverse event was unrelated to the study- patient was undergoing treatment for lung cancer.
Patient death (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — On 7/2/14 while conducting routine chart review, research staff noted that the patient passed away on 6/22/14 from a cardiac event. This adverse event was unrelated to the study- patient had a history of cardiac problems and active cocaine use.

LIMITATIONS AND CAVEATS:
This study was conducted at one VA medical center in an urban, metropolitan area. Sites can vary markedly in contextual factors; There was a large proportion of overweight patients with SMI who declined to participate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No